CLINICAL TRIAL: NCT07383974
Title: The Impact of 12 Week Retention of Nutrients on Skin and the Perception of Physical Health Status
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: W25002003
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Dietary Supplementation; Skin Health; Health Status; Antioxidants
MeSH Terms: interventions — Ascorbic Acid; Tea; Geritol; Minerals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Combination Group (Experimental)
  Interventions: Dietary Supplement: Vitamin C & Green Tea Capsules + Multivitamin & Mineral Capsules Combination
- Placebo Control Group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Combination (Matching)

INTERVENTIONS:
Dietary Supplement: Vitamin C & Green Tea Capsules + Multivitamin & Mineral Capsules Combination — Participants take a combination of active supplements-specifically, Vitamin C & Green Tea Capsules and Multivitamin & Mineral Capsules-orally twice daily.
  Arms: Supplement Combination Group
Dietary Supplement: Placebo Combination (Matching) — Participants take a matching placebo combination (identical in appearance and taste to the active supplements) orally twice daily
  Arms: Placebo Control Group

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial exploring the effects of a 12-week dietary supplement regimen on skin condition and perceived overall health status.

The study will involve 120 healthy Chinese adults aged 18 and above with low daily fruit and vegetable intake. Participants will be randomly assigned to one of two groups: one group will take a combination of Nu Skin's Vitamin C & Green Tea Capsules and Multivitamin & Mineral Capsules, while the other group will take a matching placebo.

The primary goal is to assess if the supplement combination improves skin health after 12 weeks, measured through specialized facial imaging (assessing spots, redness, evenness) and probe measurements (assessing elasticity, moisture, gloss). Secondary goals include evaluating changes in participants' self-perceived health status (via quality of life, fatigue, and digestive health questionnaires), psychological resilience, memory, and exploring a new method for measuring skin carotenoid levels.

This study is not intended to verify the approved health functions of the products but to explore the potential combined effects of antioxidant and nutritional supplementation on skin and general well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults of Asian descent aged 18 and above;
2. Daily fruit and vegetable intake < 240g (calculated based on the fruit and vegetable section of the food frequency questionnaire);
3. S3 measurement index < 30000;
4. Participants must possess basic Chinese reading comprehension and expression skills, and be able to independently complete questionnaire surveys;
5. Voluntary participation in the test and signing of the informed consent form;
6. Willingness to comply with all evaluation requirements.

Exclusion Criteria:

1. Presence of open facial skin lesions, clearly visible scars, acne marks, etc.;
2. Skin lesions, scars, or significant pigmentation on the hand measurement area;
3. Symptoms of skin disease on the face or hand measurement areas;
4. Having undergone medical aesthetic procedures within the last 6 months;
5. Participation in other clinical trials involving product use within the last 3 months;
6. Use of health supplements or nutritional supplements (e.g., vitamins, minerals) within the last 1 month;
7. Currently planning for pregnancy, pregnant, or lactating;
8. Presence of any disease under current treatment;
9. Any other health issues or chronic diseases that affect behavioral or cognitive abilities;
10. Other iatrogenic reasons identified by experts or professionals that may affect the evaluation results.

The S3 instrument refers to a Raman spectroscopy-based biophotonic scanner. The threshold for the S3 screening value is based on previously published literature, which indicated that participants with a daily fruit and vegetable intake of less than 240g had an average Raman spectroscopy biophotonic scanner score below 25,000. However, considering practical recruitment challenges, the inclusion criterion was set at < 30,000. The S3 device measures the Skin Carotenoid Index, a non-invasive biomarker reflecting skin carotenoid levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Facial Image Capture VISIA-7 | Imaging sessions are conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks)
Skin Elasticity Test Probe Cutometer | Measurements are conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks)
Skin Gloss Measurement Glossmeter | Measurements are conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).
Skin Moisture Content Corneometer | Measurements are conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks)
Skin Hemoglobin Measurement Mexameter MX18 (Courage & Khazaka, Germany) | Measurements are conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).
Skin Moisture Loss Meter Vapometer (Delfin, Finland) | Measurements are conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).
Skin Carotenoid Index | Measurements are conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).

SECONDARY OUTCOMES:
Skin Condition Survey | The scales and questionnaires are administered at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).
  This survey assesses participants' subjective perception of their skin condition over the past month. It consists of two parts: 1) The Fitzpatrick Skin Typing Questionnaire determines the participant's skin type (I-VI) based on genetic predisposition, tanning ability, and sun reaction. 2) The Skin Status Self-Assessment uses a 100mm visual analog scale for participants to rate various aspects of their skin, including photo-damage (acute and chronic), brightness, glossiness, smoothness, hydration, pore appearance, evenness, softness, elasticity, overall wrinkles, appearance, plumpness, firmness, and spots.
Physical Health and Life Status Survey | The survey is administered at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).
  This comprehensive survey evaluates participants' perceived physical health and quality of life over the past month. It incorporates five validated instruments: the SF-36 Health Survey, the Frequency of Physical Discomfort Questionnaire, the Gastrointestinal Discomfort Symptoms Questionnaire , the Population-Based Visual Fatigue Scale, and the TCM Constitution Classification and Determination Self-Assessment Table .
Psychological State and Memory Level | The assessment is conducted at T0 (baseline), T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).
  This component measures participants' subjective psychological state and memory function over the past month. It uses two main instruments: 1) The Brief Resilience Scale (BRS) assesses the ability to bounce back from stress and adversity (psychological resilience). 2) The Multifactorial Memory Questionnaire (MMQ) is divided into three subscales evaluating memory satisfaction/ability (Contentment), frequency of memory failures (Ability), and the use of compensatory strategies (Strategy).
Self-Evaluation Questionnaire | This questionnaire is administered only at follow-up visits: T4w (4 weeks), T8w (8 weeks), and T12w (12 weeks).
  This questionnaire is specifically designed for participants to subjectively evaluate the effects of the product intervention. It assesses perceived improvements in areas such as energy levels, overall health status, immune function, recovery speed from illness, quality of life, and the product's contribution to long-term health using a Likert scale.
Height and Weight Measurement BMI | Measurements are conducted at T0 (baseline, upon enrollment) and T12w (12 weeks).
  Body Mass Index (BMI) is calculated from height and weight measurements to assess weight status and changes over the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China